CLINICAL TRIAL: NCT04992910
Title: Study of the Effectiveness of Functional Electrical Stimulation Through the "Fesia Grasp" Device in the Rehabilitative Treatment of Patients With Affected Upper Limbs After a Stroke.
Brief Title: Study of the Effectiveness of "Fesia Grasp": Functional Electrical Stimulation Device for Upper Limb Rehabilitation After Stroke
Acronym: PI52021Rehab
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Collaborators: FESIA Technology (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI52021Rehab
Record Dates: First submitted 2021-07-16; First posted 2021-08-05 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Stroke; Upper Extremity Paresis
Keywords: Stroke; Upper Extremity Paresis; Functional Electrical Stimulation
MeSH Terms: conditions — Stroke; Paresis | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional Electrical Stimulation (Experimental)
  Interventions: Device: Functional electrical stimulation through medical device
- Standard Therapy (Active Comparator)
  Interventions: Other: Standard therapy

INTERVENTIONS:
Device: Functional electrical stimulation through medical device — The patient will receive a therapy with functional electrical stimulation. For this, a device called "Fesia Grasp" will be used.
  Duration: 80 min twice a week, for 6 weeks.
  Arms: Functional Electrical Stimulation
Other: Standard therapy — Physical therapy applied to the subject. Duration: 80 min twice a week, for 6 weeks.
  Arms: Standard Therapy

SUMMARY:
The purpose of this study is to evaluate the effectiveness of Fesia Grasp, a Functional Electrical Stimulation device for the rehabilitation of upper limb in post-stroke patients. Fesia Grasp rehabilitation will be compared with usual care rehabilitation of upper limb.

* Experimental group: patients will receive Fesia Grasp therapy (intensive, repetitive and functional exercises assisted by functional electrical stimulation)
* Control group - patients will receive standard care.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older subjects with hemiparesis in the upper limb after stroke, which have been referred to the Rehabilitation Unit of the Reina University Hospital.
* Unilateral paresis
* Cognitive ability to assimilate and actively participate in the protocol of evaluation and treatment

Exclusion Criteria:

* Very severe proximal spasticity: Ashworth > 3.
* Psychiatric illness (including post-stroke depression).
* Cognitive impairment.
* Inability to provide informed consent.
* Other severe medical problems.
* Severe hemi-spatial neglect or anosognosia involving the affected arm.
* Pacemakers
* Pregnant women.
* Skin ulcers.
* Peripheral neuropathies.
* Edema of the affected forearm and / or hand.
* Severe pain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-02-14 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment (FMA) scale | Change from Baseline FMA scale at 6 weeks and 3 months
  It is an index to assess the sensorimotor impairment in individuals who have had stroke. The Fugl-Meyer Assessment scale is an ordinal scale that has 3 points for each item. A zero score is given for the item if the subject cannot do the task. A score of 1 is given when the task is performed partially and a score of 2 is given when the task is performed fully. The maximun score is 66 points

SECONDARY OUTCOMES:
Medical Research Council (MRC) | Baseline; 6 weeks; 3 months
  A standardized assessment to measure muscle strength; Score range 0-5 (minimum 0, maximum 5)
Modified Ashworth Scale (MAS) | Baseline; 6 weeks; 3 months
  This scale measures resistance during passive soft-tissue stretching and is used as a simple measure of spasticity. It is single-item measures ranging from 0 to 4, where 0 indicates no increase in muscle tone and 4 indicates that the affected part is rigid in flexion or extension.
Box & Blocks Test | Baseline; 6 weeks; 3 months
  It assesses unilateral gross manual dexterity. Individuals are seated at a table, facing a rectangular box that is divided into two square compartments of equal dimension by means of a partition. One hundred and fifty, 2.5 cm, colored, wooden cubes or blocks are placed in one compartment or the other.
  The test is scored by counting the number of blocks carried over the partition from one compartment to the other during the one-minute trial period.
Motor Activity Log (MAL) | Baseline; 6 weeks; 3 months
  Semi-structured interview to assess arm function. Individuals are asked to rate Quality of Movement and Amount of Movement during 30 daily functional tasks. Target tasks include object manipulation (e.g. pen, fork, comb, and cup) as well as the use of the arm during gross motor activities (e.g. transferring to a car, steadying oneself during standing, pulling a chair into a table while sitting).
Intrinsic Motivation Inventory (IMI) | 6 weeks
  This scale is a multidimensional scale intended to assess participants subjective experience with the device (interest/enjoyment, perceived competence, effort, value/usefulness, felt pressure and tension, and perceived choice while performing a given activity). Consist of 20 item questionnaire with answers from 1 'strongly agree' to 7 'strongly disagree'.
Euroqol-5d | 6 weeks; 3 months
  Spanish version of the EuroQol-5D questionnaire (EQ-5D). It is a generic ABVD measurement instrument. The individual himself assesses his state of health, first in severity levels by five dimensions: mobility, personal care, daily activities, pain / discomfort and anxiety / depression.
Usability questionnaire specifically designed for this study | 6 weeks
  It consists of a 5 item questionnaire with five response options (Likert sacle); from Strongly agree to Strongly disagree. To evaluate the satisfaction of patients with the system and the therapy.
Adverse events | Through study completion, an average of 6 months
  Any untoward medical occurrence during the clinical trial

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Mayordomo Riera, MD, Principal Investigator — Hospital Universitario Reina Sofía
Locations (1):
- Hospital Universitario Reina Sofía, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: Yes
The results will be available for other investigators.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Once the trial is ended and the result are published in a paper.
Access Criteria: Upon request to silvia.guillen@imibic.org